CLINICAL TRIAL: NCT02554877
Title: A 12-week, Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Once Daily Pf-06291874 Administration In Adults With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: A 12-week Study To Evaluate PF-06291874 Once a Day in Adults With T2DM Inadequately Controlled On Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B4801010
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-06291874

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06291874, 30 mg (Experimental)
  Interventions: Drug: PF-06291874
- PF-06291874, 60 mg (Experimental)
  Interventions: Drug: PF-06291874
- PF-06291874, 100 mg (Experimental)
  Interventions: Drug: PF-06291874

INTERVENTIONS:
Drug: PF-06291874 — study drug to be given as an oral tablet at 30, 60 or 100 mg
  Arms: PF-06291874, 100 mg; PF-06291874, 30 mg; PF-06291874, 60 mg
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PF-06291874 is effective in the treatment T2DM

DETAILED DESCRIPTION:
This will be a randomized, double blind, stratified, placebo controlled, parallel group study conducted in T2DM subjects receiving background metformin therapy. Subjects will complete screening procedures to determine eligibility, followed by an 8 week metformin stabilization period prior to randomization. In addition, subjects taking other OADs, in combination with metformin, will undergo a washout during this period, in which non metformin OAD medications will be temporarily discontinued for the duration of the trial. Following confirmation of study eligibility criteria at randomization, subjects will be stratified into 2 groups based on the use of concomitant statin therapy. Each stratum will be randomized across treatment groups, such that the number of subjects taking concomitant statin therapy and those not taking statin therapy will be approximately balanced across treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-childbearing potential females between the ages of 18 (or the minimum country specific age of consent if >18) and 70 years, inclusive, at the screening visit (V1) with the diagnosis of T2DM;Female subjects who are not of childbearing potential
2. Subjects who have been on a stable dose of metformin either alone or in combination with one additional acceptable OAD
3. HbA1c at the Screen Visit (V1), as assessed by study specific central laboratory, is 7-11% if on metformin monotherapy; is 6.5-9.5% if on dual combination therapy (metformin plus 1)

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes;
2. Fasting plasma glucose levels >270 mg/dL (15.0 mmol/L) at the screening and run in visit, (as assessed by study specific central laboratory) confirmed by a single repeat, if deemed necessary
3. History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class III IV heart failure, or transient ischemic attack within 6 months of screening;
4. Any medical condition possibly affecting study drug absorption (eg, gastrectomy or any area of intestinal resection, active inflammatory bowel disease or pancreatic insufficiency
5. Subjects with a creatinine clearance <60 mL/min as determined by the Cockcroft Gault equation (listed below) using serum creatinine measured at screening, confirmed via a single repeat, if deemed necessary
6. Subject with a positive result for hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBc Ab) or hepatitis C virus (HCV) antibodies
7. Screening seated systolic blood pressure >160 mm Hg and/or diastolic blood pressure >105 mm Hg after at least a 5 minute rest. Blood pressure determined as the mean of triplicate measurements collected with approximately 2 minutes of rest between measurements
8. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) >470 msec; or a QRS interval >120 msec. If QTc exceeds 470 msec or QRS exceeds 120 msec, the ECG may be repeated 2 more times with an interval of 2-4 minutes between each measurement and the mean of the 3 values used to determine the subject's eligibility
9. Subjects with an arm circumference >52 cm measured at the midpoint of the length of the upper arm;
10. History (within the last 6 months) of regular alcohol consumption exceeding 14 drinks per week for men and 7 drinks a week for women. (1 drink = 5 ounces of wine (150 mL) or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor);
11. Treatment with thiazolidinediones (TZDs), or subcutaneously administered anti diabetic agents (eg, insulin, exenatide, liraglutide, pramlintide) within 6 weeks prior to V1;
12. Subjects with a known hypersensitivity or intolerance to a glucagon receptor antagonist, or known prior participation in a trial involving PF 06291874;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (32):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - National Research Institute, Los Angeles, California
  - NRC Research Institute, Orange, California
  - Sierra Clinical Research, Roseville, California
  - Encompass Clinical Research, Spring Valley, California
  - Empire Clinical Research, Upland, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Suncoast Research Group, Llc, Miami, Florida
  - QPS-MRA, LLC (Miami Research Associates), South Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - ALAS Science Clinical Research, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Clinilabs Inc., Eatontown, New Jersey
  - Pharmaceutical Research Associates, Inc., Marlton, New Jersey
  - TLB Research, Trenton, New Jersey
  - Randolph Medical Associates, Asheboro, North Carolina
  - High Point Clinical Trials Center, LLC, High Point, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Aventiv Research, Columbus, Ohio
  - Juno Research, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Juno Research, LLC, Katy, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC, Schertz, Texas
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
- Canada (6):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - LMC Clinical Research Inc. (Thornhill), Thornhill, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Manna Research Inc., Lévis, Quebec
  - Omnispec Clinical Research, Inc., Mirabel, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4801010

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Four (4) tablets of placebo matched to PF-06291874 and at least 1 stable dose of open label metformin were orally administered with a standard morning meal once daily for 12 weeks.
- PF-06291874 30 mg: Two (2) placebo tablets, one 5-mg and one 25-mg of PF-06291874 tablets and at least 1 stable dose of open label metformin were orally administered with a standard morning meal once daily for 12 weeks.
- PF-06291874 60 mg: Two (2) 5-mg and two 25-mg of PF-06291874 tablets and at least 1 stable dose of open label metformin were orally administered with a standard morning meal once daily for 12 weeks.
- PF-06291874 100 mg: Four (4) 25-mg of PF-06291874 tablets and at least 1 stable dose of open label metformin were orally administered with a standard morning meal once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Started | 51 | 51 | 52 | 52
Completed | 39 | 44 | 46 | 45
Not Completed | 12 | 7 | 6 | 7
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2
Not completed — Did not meet entrance criteria | 0 | 0 | 1 | 0
Not completed — No longer met eligibility criteria | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 1 | 1 | 0
Not completed — Other | 1 | 3 | 0 | 3
Not completed — Insufficient clinical response | 4 | 0 | 0 | 0
Not completed — No longer willing to participate | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg | Total
Number analyzed (Participants) | 51 | 51 | 52 | 52 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (6.3) | 58.1 (6.9) | 57.1 (7.1) | 57.4 (7.9) | 57.3 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 24 | 21 | 87
  Male | 29 | 31 | 28 | 31 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) (%) at Week 12 as Compared to Placebo
Description: HbA1c was a form of hemoglobin which was measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Baseline was defined as the last pre-dose measurement prior to first double blind dosing for the study.
Time Frame: Baseline, Week 12
Population: All participants randomized and who received at least 1 dose of randomized treatment, participants were assigned to the randomized treatment regardless of what treatment was received.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 39 | 44 | 46 | 45
percentage of HbA1c | 0.18 (0.834) | -0.68 (0.778) | -0.91 (0.765) | -0.92 (0.809)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Two (2)-sided p-values were from mixed model for repeated measurements (MMRM) with baseline value, time (study day), treatment group, time by treatment interaction as fixed effects and an unstructured correlation matrix; LS Mean difference from placebo = -0.91, 95% CI 2-sided [-1.34 to -0.48], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean difference from placebo = -1.16, 95% CI 2-sided [-1.59 to -0.73], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean difference from placebo = -1.17, 95% CI 2-sided [-1.60 to -0.74], Standard Error of Mean 0.16

2. Secondary Outcome: Change From Baseline in HbA1c (%) at Weeks 2, 4, and 8
Description: HbA1c was a form of hemoglobin which was measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Baseline was defined as the last pre-dose measurement prior to first double blind dosing for the study. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8
Population: All participants randomized and who received at least 1 dose of randomized treatment, participants were assigned to the randomized treatment regardless of what treatment was received.n represented the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
percentage of HbA1c
  Week 2 HbA1c(%)Change from Baseline(n=46,48,48,47) | 0.10 (0.363) | -0.30 (0.383) | -0.30 (0.341) | -0.31 (0.260)
  Week 4 HbA1c(%)Change from Baseline(n=45,47,47,47) | 0.12 (0.426) | -0.53 (0.546) | -0.57 (0.444) | -0.49 (0.371)
  Week 8 HbA1c(%)Change from Baseline(n=40,45,47,45) | 0.15 (0.653) | -0.65 (0.617) | -0.90 (0.612) | -0.82 (0.512)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two (2)-sided p-values were from analysis of covariance (ANCOVA) model with baseline value and treatment group as fixed effects; Least squares mean (LS mean) difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.39, 95% CI 2-sided [-0.52 to -0.26], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.39, 95% CI 2-sided [-0.52 to -0.26], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.44, 95% CI 2-sided [-0.57 to -0.30], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.59, 95% CI 2-sided [-0.76 to -0.42], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.63, 95% CI 2-sided [-0.80 to -0.46], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.62, 95% CI 2-sided [-0.79 to -0.46], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.71, 95% CI 2-sided [-0.93 to -0.49], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.96, 95% CI 2-sided [-1.17 to -0.74], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference from placebo adjusted for baseline values was derived from the ANCOVA model; LS Mean difference from placebo = -0.98, 95% CI 2-sided [-1.20 to -0.76], Standard Error of Mean 0.11

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Weeks 2, 4, 8, and 12
Description: Fasting plasma glucose response changed from baseline at Weeks 2,4,8 and 12. Baseline was defined as the average of the measurements obtained during Day 14 visit window and Day 1 pre-dose measurement. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2,4,8 and 12
Population: All participants randomized and who had received at least 1 dose of randomized treatment. n represented the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
mg/dL
  Week 2 Change from Baseline(n=49,48,48,47) | 11.0 (28.5) | -25.2 (26.95) | -32.4 (35.31) | -32.5 (32.26)
  Week 4 Change from Baseline(n=45,47,47,47) | 3.4 (29.22) | -26.8 (29.68) | -34.7 (39.15) | -30.9 (32.55)
  Week 8 Change from Baseline(n=39,44,47,45) | -1.8 (42.57) | -19.9 (35.93) | -35.4 (32.5) | -31.8 (26.57)
  Week 12 Change from Baseline(n=39,43,46,45) | -0.6 (31.64) | -18.5 (30.19) | -32.8 (35.24) | -31.9 (35.56)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Two (2)-sided p-values were from MMRM with baseline value, time (study day), treatment group, time by treatment interaction as fixed effects and an unstructured correlation matrix; LS Mean difference from placebo = -37.83, 95% CI 2-sided [-47.96 to -27.70], Standard Error of Mean 5.13
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -44.85, 95% CI 2-sided [-54.98 to -34.72], Standard Error of Mean 5.13
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -48.59, 95% CI 2-sided [-58.81 to -38.37], Standard Error of Mean 5.18
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -30.63, 95% CI 2-sided [-42.52 to -18.74], Standard Error of Mean 6.03
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -39.24, 95% CI 2-sided [-51.13 to -27.35], Standard Error of Mean 6.03
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -38.30, 95% CI 2-sided [-50.22 to -26.38], Standard Error of Mean 6.04
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -19.47, 95% CI 2-sided [-31.88 to -7.05], Standard Error of Mean 6.29
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -36.98, 95% CI 2-sided [-49.27 to -24.69], Standard Error of Mean 6.23
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -35.14, 95% CI 2-sided [-47.55 to -22.72], Standard Error of Mean 6.29
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -19.77, 95% CI 2-sided [-31.81 to -7.73], Standard Error of Mean 6.10
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -35.26, 95% CI 2-sided [-47.17 to -23.35], Standard Error of Mean 6.03
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -36.44, 95% CI 2-sided [-48.43 to -24.46], Standard Error of Mean 6.07

4. Secondary Outcome: Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c) <7% as Well as <6.5% at Week 12.
Description: HbA1c was a form of hemoglobin which was measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % (percentage of participants)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 39 | 44 | 46 | 45
% (percentage of participants)
  HbA1c <6.5% | 5.13 [0.63 to 17.32] | 11.36 [3.79 to 24.56] | 13.04 [4.94 to 26.26] | 22.22 [11.20 to 37.09]
  HbA1c <7% | 15.38 [5.86 to 30.53] | 29.55 [16.76 to 45.20] | 34.78 [21.35 to 50.25] | 55.56 [40.00 to 70.36]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<7%); Test type: Superiority or Other; p = 0.0059, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Odds Ratio (OR) = 6.057, 95% CI 2-sided [1.68 to 21.82]
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<7%); Test type: Superiority or Other; p = 0.0008, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Odds Ratio (OR) = 8.927, 95% CI 2-sided [2.49 to 31.96]
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<7%); Test type: Superiority or Other; p < 0.0001, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Odds Ratio (OR) = 15.116, 95% CI 2-sided [4.34 to 52.67]
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<6.5%); Test type: Superiority or Other; p = 0.1532, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Odds Ratio (OR) = 3.340, 95% CI 2-sided [0.64 to 17.47]
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<6.5%); Test type: Superiority or Other; p = 0.0826, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Risk Ratio (RR) = 4.198, 95% CI 2-sided [0.83 to 21.22]
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12 (HbA1C<6.5%); Test type: Superiority or Other; p = 0.0272, Regression, Logistic — P-value was derived from the logistic regression model with treatment (categorical) and baseline HbA1c as covariate; Odds Ratio (OR) = 5.588, 95% CI 2-sided [1.21 to 25.73]

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The total number of participants with laboratory test abnormalities (without regard to baseline abnormality) was assessed. Clinical laboratory tests included hematology, chemistry, urinalysis, and some other tests.
Time Frame: Baseline up to 98 days
Population: The safety analysis set was used, which defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 49 | 51 | 50
participants | 49 | 42 | 40 | 38

6. Secondary Outcome: Number of Participants With Change From Baseline and Absolute Values in 12-lead Electrocardiograms (ECGs) Meeting Categorical Summarization Criteria
Description: ECG criteria of potential clinical concern were 1), time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval): >=140 milliseconds (msec); >=50% increase from baseline; 2), the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval): >=300 msec; >=25 percent (%) increase when baseline >200 msec; or increase >=50% when baseline less than or equal to (<=)200 msec; 3), time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec, >=500 msec; increase from baseline >=30 - <60, >=60 msec.
Time Frame: Baseline up to Day 98
Population: The safety analysis set was used, which defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 48 | 50 | 50
participants
  Maximum PR interval >=300 msec | 0 | 0 | 0 | 0
  Maximum QRS interval >=140 msec | 0 | 0 | 0 | 1
  Maximum QTcF interval 450-<480 msec | 4 | 4 | 2 | 2
  Maximum PR interval increase >=25%/50% | 0 | 0 | 1 | 1
  Maximum QRS complex increase >=50% | 1 | 0 | 0 | 0
  Maximum QTcF interval increase 30<=-<60 msec | 1 | 0 | 3 | 5
  Maximum QTcF interval increase >=60 msec | 0 | 1 | 0 | 0
  Maximum QTcF interval 480-<500 msec | 0 | 0 | 0 | 0
  Maximum QTcF interval >=500 msec | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Categorical Summarization Criteria
Description: Vital signs included seated supine systolic and diastolic blood pressure (BP) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from baseline, diastolic <50 mm Hg; 2), pulse rate <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: Baseline up to Day 98
Population: The safety analysis set was used, which defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 49 | 51 | 50
participants
  Sitting SBP <90 mm Hg | 1 | 0 | 0 | 0
  Sitting DBP <50mm Hg | 1 | 0 | 0 | 0
  Sitting Pulse Rate <40 bpm | 0 | 0 | 0 | 0
  Sitting Pulse Rate >120 bpm | 0 | 0 | 0 | 0
  Increase: Sitting SBP >=30 mm Hg | 0 | 3 | 1 | 4
  Increase: Sitting Systolic BP >=20 mm Hg | 0 | 1 | 0 | 3
  Decrease: Sitting SBP >=30 mm Hg | 1 | 2 | 1 | 0
  Decrease: Sitting SBP >=20 mm Hg | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Hypoglycemic Adverse Events (HAEs).
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a study drug; the event need not necessarily have a causal relationship with the treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reasons: death; life threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. An HAE was identified by characteristic symptoms or blood glucose levels. Any events occurring following start of treatment (defined as blinded therapy, including single blind placebo administration on Day 14) or increasing in severity were counted as treatment emergent AE.
Time Frame: Baseline up to Day 119
Population: The safety analysis set was used, which defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
participants
  AEs | 22 | 20 | 18 | 27
  SAEs | 2 | 1 | 0 | 2
  HAEs | 5 | 1 | 1 | 2

9. Secondary Outcome: Percent Changes From Baseline for Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Weeks 2, 4, 8 and 12
Description: Fasting low density lipoprotein-cholesterol (LDL-C) percent change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) at Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: All participants randomized and who received at least 1 dose of randomized treatment, participants were assigned to the randomized treatment regardless of what treatment was received. n represented the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
% (percent change)
  Week 2 Percent Change from Baseline(n=49,47,48,47) | 0.68 (16.301) | -1.41 (17.832) | -0.64 (17.154) | 2.16 (16.846)
  Week 4 Percent Change from Baseline(n=45,47,47,47) | 3.29 (18.485) | 0.46 (12.752) | -0.62 (18.522) | -2.07 (15.170)
  Week 8 Percent Change from Baseline(n=40,45,47,45) | 5.31 (21.244) | 2.17 (15.503) | 1.32 (17.448) | 1.92 (17.030)
  Week12 Percent Change from Baseline(n=39,43,46,45) | 0.13 (18.680) | 1.77 (17.278) | 4.20 (18.315) | 1.16 (19.061)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.7618, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -1.03, 90% CI 2-sided [-6.66 to 4.59], Standard Error of Mean 3.40
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.8489, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -0.65, 90% CI 2-sided [-6.25 to 4.96], Standard Error of Mean 3.39
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.4699, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 2.47, 90% CI 2-sided [-3.17 to 8.12], Standard Error of Mean 3.42
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.4979, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -2.22, 90% CI 2-sided [-7.63 to 3.19], Standard Error of Mean 3.27
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.2927, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -3.45, 90% CI 2-sided [-8.85 to 1.95], Standard Error of Mean 3.27
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.1430, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -4.83, 90% CI 2-sided [-10.26 to 0.60], Standard Error of Mean 3.28
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.7373, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -1.25, 90% CI 2-sided [-7.42 to 4.92], Standard Error of Mean 3.73
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.5075, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -2.46, 90% CI 2-sided [-8.57 to 3.66], Standard Error of Mean 3.70
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.6295, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -1.81, 90% CI 2-sided [-7.99 to 4.37], Standard Error of Mean 3.74
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.4266, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.15, 90% CI 2-sided [-3.39 to 9.69], Standard Error of Mean 3.95
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.2038, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 4.96, 90% CI 2-sided [-1.47 to 11.40], Standard Error of Mean 3.89
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.5592, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 2.29, 90% CI 2-sided [-4.19 to 8.78], Standard Error of Mean 3.92

10. Secondary Outcome: Percent Changes From Baseline for Triglycerides at Weeks 2, 4, 8 and 12
Description: Triglycerides percent change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) at Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days. Triglycerides MMRM was not appropriate as the data were very skewed and not normally distributed, therefore per SAP non-parametric analysis were reported, presenting medians and CIs for medians, instead. If the data had many outliers even after the log transformation the following non parametric analysis was presented instead of the MMRM. An outlier was defined as any data point falling outside of 3.5 x standard deviations the median.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 9
Measure: Median (Full Range); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
% (percent change)
  Week 2 Percent Change from Baseline(n=49,48,48,47) | 5.45 [-56.7 to 126.3] | 10.55 [-44.0 to 138.5] | 8.32 [-32.6 to 189.0] | 22.58 [-37.5 to 144.7]
  Week 4 Percent Change from Baseline(n=44,47,47,47) | 3.74 [-59.0 to 224.1] | 6.45 [-48.2 to 121.4] | 6.67 [-44.8 to 169.8] | 1.18 [-35.7 to 107.2]
  Week 8 Percent Change from Baseline(n=40,45,47,45) | 6.72 [-37.7 to 155.2] | 5.08 [-36.9 to 103.9] | 2.13 [-52.1 to 178.1] | 9.47 [-49.3 to 140.0]
  Week12 Percent Change from Baseline(n=39,44,46,45) | -0.72 [-38.4 to 154.0] | 7.13 [-47.7 to 186.7] | -1.85 [-48.0 to 147.8] | 5.26 [-47.9 to 112.6]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; Median Difference (Net) = 5.09, 90% CI 2-sided [-5.86 to 16.05]
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; Median Difference (Net) = 2.86, 90% CI 2-sided [-9.76 to 15.48]
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; Median Difference (Net) = 17.13, 90% CI 2-sided [3.91 to 30.34]
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; Median Difference (Net) = 2.71, 90% CI 2-sided [-10.80 to 16.22]
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; Median Difference (Net) = 2.92, 90% CI 2-sided [-10.61 to 16.45]
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; Median Difference (Net) = -2.57, 90% CI 2-sided [-15.08 to 9.94]
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; Median Difference (Net) = -1.63, 90% CI 2-sided [-16.29 to 13.03]
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; Median Difference (Net) = -4.59, 90% CI 2-sided [-20.40 to 11.22]
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; Median Difference (Net) = 2.75, 90% CI 2-sided [-13.66 to 19.16]
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; Median Difference (Net) = 7.86, 90% CI 2-sided [-3.30 to 19.02]
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; Median Difference (Net) = -1.13, 90% CI 2-sided [-16.13 to 13.87]
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; Median Difference (Net) = 5.99, 90% CI 2-sided [-7.07 to 19.04]

11. Secondary Outcome: Percent Changes From Baseline for Total Cholesterol at Weeks 2, 4, 8 and 12
Description: Total cholesterol percent change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) on Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
% (percent change)
  Week 2 Percent Change from Baseline(n=49,48,48,47) | 0.16 (11.863) | 0.39 (12.606) | 1.02 (12.058) | 4.05 (13.900)
  Week 4 Percent Change from Baseline(n=44,47,47,47) | 2.65 (14.642) | 1.69 (8.763) | 0.36 (13.732) | 0.44 (11.674)
  Week 8 Percent Change from Baseline(n=40,45,47,45) | 3.30 (14.354) | 1.53 (10.569) | -0.11 (12.692) | 2.77 (10.860)
  Week12 Percent Change from Baseline(n=39,44,46,45) | -0.87 (13.238) | 2.28 (12.260) | 3.00 (13.952) | 2.03 (13.986)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.6800, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.04, 90% CI 2-sided [-3.12 to 5.20], Standard Error of Mean 2.52
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.5150, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.64, 90% CI 2-sided [-2.52 to 5.80], Standard Error of Mean 2.52
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.0676, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 4.66, 90% CI 2-sided [0.47 to 8.85], Standard Error of Mean 2.53
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.8021, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -0.62, 90% CI 2-sided [-4.73 to 3.48], Standard Error of Mean 2.48
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.4346, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -1.95, 90% CI 2-sided [-6.06 to 2.16], Standard Error of Mean 2.49
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.4173, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -2.03, 90% CI 2-sided [-6.15 to 2.09], Standard Error of Mean 2.49
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.7036, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -0.98, 90% CI 2-sided [-5.21 to 3.26], Standard Error of Mean 2.56
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.2993, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -2.64, 90% CI 2-sided [-6.84 to 1.56], Standard Error of Mean 2.54
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.9751, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.08, 90% CI 2-sided [-4.16 to 4.32], Standard Error of Mean 2.57
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.1408, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 4.23, 90% CI 2-sided [-0.50 to 8.96], Standard Error of Mean 2.86
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0986, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 4.70, 90% CI 2-sided [0.02 to 9.38], Standard Error of Mean 2.83
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.1851, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.79, 90% CI 2-sided [-0.92 to 8.50], Standard Error of Mean 2.85

12. Secondary Outcome: Percent Changes From Baseline for High Density Lipoprotein-Cholesterol (HDL-C) at Weeks 2, 4, 8 and 12
Description: High density lipoprotein-cholesterol (HDL-C) percent change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) at Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
% (percent change)
  Week 2 Percent Change from Baseline(n=49,48,48,47) | -0.14 (8.086) | 0.08 (9.345) | 2.60 (10.739) | 8.13 (13.554)
  Week 4 Percent Change from Baseline(n=44,47,47,47) | 0.51 (11.391) | 0.79 (10.626) | 3.98 (14.288) | 8.16 (11.776)
  Week 8 Percent Change from Baseline(n=40,45,47,45) | -1.91 (11.736) | 1.24 (10.292) | 2.15 (10.724) | 7.71 (13.768)
  Week12 Percent Change from Baseline(n=39,44,46,45) | -2.62 (13.237) | 3.65 (12.889) | 4.51 (10.598) | 7.57 (15.226)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.8559, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.39, 90% CI 2-sided [-3.19 to 3.98], Standard Error of Mean 2.17
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.1729, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 2.97, 90% CI 2-sided [-0.62 to 6.55], Standard Error of Mean 2.17
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 8.45, 90% CI 2-sided [4.84 to 12.06], Standard Error of Mean 2.18
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.8837, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.37, 90% CI 2-sided [-3.85 to 4.59], Standard Error of Mean 2.55
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.1573, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.62, 90% CI 2-sided [-0.60 to 7.84], Standard Error of Mean 2.55
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 7.88, 90% CI 2-sided [3.65 to 12.11], Standard Error of Mean 2.56
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.1538, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.59, 90% CI 2-sided [-0.55 to 7.73], Standard Error of Mean 2.51
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.0789, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 4.39, 90% CI 2-sided [0.28 to 8.49], Standard Error of Mean 2.48
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 10.14, 90% CI 2-sided [5.98 to 14.30], Standard Error of Mean 2.51
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0132, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 6.96, 90% CI 2-sided [2.36 to 11.56], Standard Error of Mean 2.78
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0079, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 7.41, 90% CI 2-sided [2.85 to 11.96], Standard Error of Mean 2.75
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 10.83, 90% CI 2-sided [6.24 to 15.42], Standard Error of Mean 2.77

13. Secondary Outcome: Percent Changes From Baseline for Non-High Density Lipoprotein (HDL) Cholesterol at Weeks 2, 4, 8 and 12
Description: Non-HDL-C percent change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) on Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
% (percent change)
  Week 2 Percent Change from Baseline(n=49,48,48,47) | 0.51 (16.195) | 1.00 (16.675) | 0.63 (14.870) | 2.73 (18.427)
  Week 4 Percent Change from Baseline(n=44,47,47,47) | 4.18 (21.486) | 1.88 (11.961) | -0.47 (17.972) | -2.40 (13.877)
  Week 8 Percent Change from Baseline(n=40,45,47,45) | 5.24 (19.222) | 1.76 (14.128) | -0.52 (16.014) | 0.88 (13.765)
  Week12 Percent Change from Baseline(n=39,44,46,45) | -0.48 (16.711) | 2.09 (16.451) | 2.67 (18.098) | -0.25 (17.666)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.6597, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.46, 90% CI 2-sided [-4.01 to 6.92], Standard Error of Mean 3.31
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.7583, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.02, 90% CI 2-sided [-4.45 to 6.49], Standard Error of Mean 3.31
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.3516, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.11, 90% CI 2-sided [-2.39 to 8.61], Standard Error of Mean 3.33
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.5877, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -1.83, 90% CI 2-sided [-7.42 to 3.75], Standard Error of Mean 3.38
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.2016, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -4.33, 90% CI 2-sided [-9.92 to 1.26], Standard Error of Mean 3.38
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.0568, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -6.49, 90% CI 2-sided [-12.08 to -0.89], Standard Error of Mean 3.39
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.3827, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -2.94, 90% CI 2-sided [-8.48 to 2.61], Standard Error of Mean 3.36
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.1126, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -5.31, 90% CI 2-sided [-10.81 to 0.20], Standard Error of Mean 3.33
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.2160, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = -4.17, 90% CI 2-sided [-9.73 to 1.38], Standard Error of Mean 3.36
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.3443, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.54, 90% CI 2-sided [-2.64 to 9.72], Standard Error of Mean 3.74
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.3031, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 3.82, 90% CI 2-sided [-2.30 to 9.94], Standard Error of Mean 3.70
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.8129, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.88, 90% CI 2-sided [-5.27 to 7.04], Standard Error of Mean 3.72

14. Secondary Outcome: Changes From Baseline in Body Weight at Weeks 2, 4, 8, and 12.
Description: The body weight change from baseline (defined as the mean of Day 14 and Day 1 pre-dose) at Weeks 2,4,8 and 12. n represented the available number of participants for analysis at post-baseline days.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
kg
  Week 2 Change from Baseline(n=49,48,48,47) | -0.15 (1.347) | 0.15 (1.234) | -0.15 (1.253) | 0.65 (3.342)
  Week 4 Change from Baseline(n=45,47,47,47) | -0.76 (3.302) | 0.55 (1.231) | 0.28 (1.219) | 0.56 (2.925)
  Week 8 Change from Baseline(n=41,45,47,45) | -0.61 (1.517) | 0.44 (1.694) | 0.26 (1.775) | 0.55 (2.786)
  Week 12 Change from Baseline(n=39,44,46,45) | -0.79 (1.892) | 0.49 (2.119) | 0.31 (2.135) | 0.41 (3.216)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.4020, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.34, 90% CI 2-sided [-0.33 to 1.01], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.8789, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.06, 90% CI 2-sided [-0.61 to 0.73], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 2; Test type: Superiority or Other; p = 0.0345, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.87, 90% CI 2-sided [0.19 to 1.54], Standard Error of Mean 0.41
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.0087, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.28, 90% CI 2-sided [0.48 to 2.08], Standard Error of Mean 0.48
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.0268, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.08, 90% CI 2-sided [0.28 to 1.88], Standard Error of Mean 0.48
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 4; Test type: Superiority or Other; p = 0.0047, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.39, 90% CI 2-sided [0.58 to 2.19], Standard Error of Mean 0.49
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.07, 90% CI 2-sided [0.38 to 1.76], Standard Error of Mean 0.42
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.0220, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.97, 90% CI 2-sided [0.27 to 1.66], Standard Error of Mean 0.42
Statistical Analysis 9: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 8; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.31, 90% CI 2-sided [0.62 to 2.01], Standard Error of Mean 0.42
Statistical Analysis 10: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.41, 90% CI 2-sided [0.56 to 2.26], Standard Error of Mean 0.51
Statistical Analysis 11: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0225, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.18, 90% CI 2-sided [0.33 to 2.02], Standard Error of Mean 0.51
Statistical Analysis 12: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the reference and each of the active doses was the test for Week 12; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.40, 90% CI 2-sided [0.55 to 2.25], Standard Error of Mean 0.51
Statistical Analysis 13: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 2. The readings with residual greater than 3.5 times of its standard derivation were excluded from the presentation. (Excluding outliers); Test type: Superiority or Other; p = 0.2391, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.30, 90% CI 2-sided [-0.12 to 0.73], Standard Error of Mean 0.26
Statistical Analysis 14: Comparison: Placebo vs PF-06291874 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.9912, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.00, 90% CI 2-sided [-0.42 to 0.43], Standard Error of Mean 0.26
Statistical Analysis 15: Comparison: Placebo vs PF-06291874 100 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1930, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.34, 90% CI 2-sided [-0.09 to 0.77], Standard Error of Mean 0.26
Statistical Analysis 16: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 4. The readings with residual greater than 3.5 times of its standard derivation were excluded from the presentation. (Excluding outliers); Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.80, 90% CI 2-sided [0.35 to 1.25], Standard Error of Mean 0.27
Statistical Analysis 17: Comparison: Placebo vs PF-06291874 60 mg; Placebo was the reference and each of the active doses was the test for Week 4. The readings with residual greater than 3.5 times of its standard derivation were excluded from the presentation.(Excluding outliers); Test type: Superiority or Other; p = 0.0394, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.57, 90% CI 2-sided [0.12 to 1.02], Standard Error of Mean 0.27
Statistical Analysis 18: Comparison: Placebo vs PF-06291874 100 mg; [analysis description as in outcome 14, analysis 17]; Test type: Superiority or Other; p = 0.0862, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.48, 90% CI 2-sided [0.02 to 0.93], Standard Error of Mean 0.28
Statistical Analysis 19: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 8. The readings with residual greater than 3.5 times of its standard derivation were excluded from the presentation.(Excluding outliers); Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.05, 90% CI 2-sided [0.48 to 1.61], Standard Error of Mean 0.34
Statistical Analysis 20: Comparison: Placebo vs PF-06291874 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0068, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.92, 90% CI 2-sided [0.37 to 1.48], Standard Error of Mean 0.34
Statistical Analysis 21: Comparison: Placebo vs PF-06291874 100 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0132, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.86, 90% CI 2-sided [0.29 to 1.42], Standard Error of Mean 0.34
Statistical Analysis 22: Comparison: Placebo vs PF-06291874 30 mg; Placebo was the reference and each of the active doses was the test for Week 12. The readings with residual greater than 3.5 times of its standard derivation were excluded from the presentation.(Excluding outliers); Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.39, 90% CI 2-sided [0.65 to 2.14], Standard Error of Mean 0.45
Statistical Analysis 23: Comparison: Placebo vs PF-06291874 60 mg; [analysis description as in outcome 14, analysis 22]; Test type: Superiority or Other; p = 0.0115, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 1.15, 90% CI 2-sided [0.40 to 1.89], Standard Error of Mean 0.45
Statistical Analysis 24: Comparison: Placebo vs PF-06291874 100 mg; [analysis description as in outcome 14, analysis 22]; Test type: Superiority or Other; p = 0.0344, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference from placebo = 0.97, 90% CI 2-sided [0.22 to 1.72], Standard Error of Mean 0.45

ADVERSE EVENTS:
Time Frame: Baseline up to Day 119
Description: The same event might have appeared as both an AE and an SAE. However, what is presented are distinct events. An event might have been categorized as serious in 1 participant and as non-serious in another participant, or 1 participant might have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | PF-06291874 30 mg | PF-06291874 60 mg | PF-06291874 100 mg
Serious Adverse Events (participants affected / at risk) | 2/51 | 1/51 | 0/52 | 2/52
Other Adverse Events (participants affected / at risk) | 6/51 | 5/51 | 2/52 | 7/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | PF-06291874 30 mg (N=51) | PF-06291874 60 mg (N=52) | PF-06291874 100 mg (N=52)
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | PF-06291874 30 mg (N=51) | PF-06291874 60 mg (N=52) | PF-06291874 100 mg (N=52)
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.